CLINICAL TRIAL: NCT02652013
Title: Evaluation and Neural Basis of Communication in Patients With Multiple Sclerosis
Acronym: COGNISEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: Rennes University Hospital (Other); University Hospital, Angers (Other Government); Université Européenne de Bretagne (Other)
Responsible Party: Principal Investigator, Philippe Gallien, Medical Doctor HDR, Pôle Saint Hélier
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2015-A00624-45
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis; Social Cognition; Neuropsychology; Psychological Therory; Theory of Mind
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40 patients with multiple sclerosis (Experimental): The study sample will consist of 40 patients with multiple sclerosis. MS patients and control subjects will be recruited on the Rennes (Centre Hospitalier Universitaire and Pôle de Médecine Physique et de Réadaptation Saint-Hélier) and Angers sites (Centre Hospitalier Universitaire) participating in COGNISEP project
  Interventions: Other: cognitive evaluation
- 40 healthy subjects (Other): All the performance of the 40 MS patients will be compared to 40 control subjects matched in age, gender and sociocultural level. Subjects with a history of neurological and psychiatric condition or substance abuse will be excluded from the study. Control subjects will receive an honorary as a token for their time.
  Interventions: Other: cognitive evaluation

INTERVENTIONS:
Other: cognitive evaluation

SUMMARY:
Multiple sclerosis (MS) progressively leads to an increasing level of disability. That's why individuals faced with this chronic disease whose progression is unpredictable have to mobilize all their available resources. As a result, management of interpersonal relationships appears to be a key issue in adjustment to situations.

Although knowledge on cognitive abnormalities in MS has been growing in recent years, there is a lack of research about social behaviour regulation skills. The few studies conducted in this field are mainly interested in emotional processing (emotional facial recognition and empathy) and skills mentalizing (theory of mind) that appear disturbed in MS.

While some recent studies touch on the issue of the contextual analysis of language (that is to say, the social use of language) in MS, their assessment on a wide range of pragamtic skills has never been studied. However, the pragmatic aspects of language are known to play a major role in social adjustment.

This project has three main objectives : (1) to increase general knowledge of deficits in communication and in social cognition in patients with MS, (2) to propose new leads for the evaluation of these disorders and (3) to contribute to increasing knowledge of neural basis of communication and social cognition.

In order to address those objectives, the assessment will be focused on many various pragmatics skills : conversation, indirect language comprehension (indirect questions, idiomatic expressions, sarcasm) and metapragmatic knowledge in a population of 40 RR-MS patients. Those patients' performances will be compared to a group of healthy matched control subjects, potential relationships between pragmatic abilities, other aspects of social cognition (theory of mind and processing of emotional stimuli), cognitive functioning, psycho-behavioural aspects and the characteristics of the disease will be explore.

Social cognition tasks have been selected for their dynamic and ecologic aspects in order to match natural social interaction.

Finally, communication consideration, cognitive and cerebral skills of patients with MS will contribute to increasing knowledge of the neural basis of social cognition.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Relapsing-remitting form as defined by the Mc Donald's Committee criteria (2005).
* EDSS between 0 and 5.5, out of relapses
* French mother tongue or having been schooled in France
* No disorders of formal language comprehension
* Not having participated to a similar protocol within the 9 months preceding the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
conversation test | fist day of the assessment
  The objective of this task is to assess the verbal communication skills of MS patients in a 10-minute natural conversation (various conversation topics appropriated to the participant's age will be inserted in the conversation). Different performance indexes will be analyzed in this task: amount of verbal exchanges between both interlocutors (number of turn-taking and statements), adjustment to the examiner's requests, topic changes and topic continuity. With the use of the validated observation grid ("protocole Montréal d'évaluation de la Communication"), it will be possible to measure the frequency of occurrence or intensity of communicative behaviours
indirect langage comprehension | second day of the assesment
  This computer-based task assesses the MS patients' ability to understand indirect statements. Three forms of indirect language will be tested in this protocol: indirect requests, idiomatic expressions and sarcasms (12 items per language forms). Each item consists of a story (3 pictures with an audio-recorded text) where at least 2 characters appear in everyday life situations. The participant has to choose the end of the story from the four options (pragmatic evaluation) and to justify his/her answer (metapragmatic evaluation). The performance indexes used are the total number of correct answers, the total number of correct answers by linguistic form and the number of central justifications by correct answer, showing metapragmatic knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, doctor, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pôle Saint Hélier, Rennes, Brittany Region, France